CLINICAL TRIAL: NCT05269225
Title: Organic Diet in Pregnancy and Risk Markers of Health Effects
Brief Title: Organic Diet in Pregnancy and Risk Markers of Health Effects (The OrgDiet Project)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Per Ole Iversen, MD (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor-Investigator, Per Ole Iversen, MD, Professor, University of Oslo
Organization: University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 304336
Record Dates: First submitted 2022-02-01; First posted 2022-03-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Organic diet (Experimental): Consuming organic food from the start of 2nd trimester and until gestational week 37.
  Interventions: Other: Organic diet
- Conventional diet (Placebo Comparator): Consuming conventional food throughout the whole pregnancy.
  Interventions: Other: Conventional diet

INTERVENTIONS:
Other: Organic diet — Organically produced foods.
  Arms: Organic diet
Other: Conventional diet — Conventionally produced foods.
  Other Names: Control
  Arms: Conventional diet

SUMMARY:
The OrgDiet project is a two-armed (1:1), open, intention-to-treat randomized controlled trial. The aim is to examine effects of consumption of organic foods (intervention group) vs. conventional foods (control group) during pregnancy in both mother and child. About 100 participants will be included and the participants will be followed until the children are two years old. Both groups will also be recommended to eat according to the dietary guidelines of the Directory of Health in Norway.

ELIGIBILITY:
Inclusion Criteria:

* Nulli- or multipara pregnant in first trimester

Exclusion Criteria:

* Consuming an organic diet regularly
* Using medication regularly that might interfere with study adherence or - outcomes
* Diagnosed with a chronic disorder or cancer
* Having a food allergy or intolerance

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only pregnant women will be included
Enrollment: 100 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal urinary excretion level of dialkylphosphates | 2.5 years
  The difference in maternal urinary excretion level of these pesticides at the end of intervention (gestational week 37) between the intervention group and the control group, measured at baseline (gestational week 12-14), and at several occasions until 2 years after the birth of the baby.

SECONDARY OUTCOMES:
Blood concentration of cholesterol | 2.5 years
  The difference in blood concentration of cholesterol at the end of intervention (gestational week 37) between the intervention group and the control group, measured at baseline (gestational week 12-14), and at several occasions until 2 years after the birth of the baby.
Abundance and species-types of gut microbiota (e.g. staphylococci and enterobacter) sampled from stool samples | 2.5 years
  The difference in microbiota species-types and abundance (using 16S rRNA amplicon sequencing) in stool samples between the intervention group and the control group, measured at baseline (gestational week 12-14), and at several occasions until 2 years after the birth of the baby.
DNA methylation patterns in leucocytes as a marker of altered epigenetic programming | 2.5 years
  DNA methylation will be investigated on DNA isolated from leukocytes. Degree of DNA methylation will be analyzed at a genome-wide scale using Illumina Infinium EPIC bead chip array (or similar methods, depending on the cost-benefit consideration at the time). The DNA methylation data will be normalized, and presented as beta-values ranging from 0-1. The outcome measure in the study is intra-individual DNA methylation changes during the study-period, measured as changes in the beta-value, between the intervention group and the control group, measured at baseline (gestational week 12-14), and at several occasions until 2 years after the birth of the baby.
Child body weight | 2 years
  The difference in child body weight (kg) between the intervention group and the control group, measured at baseline (birth), and at several occasions until 2 years after the birth of the baby.
Child urinary excretion level of dialkylphosphates | 2 years
  The difference in child urinary excretion level of dialkylphosphates between the intervention group and the control group, measured at several occasions until 2 years after the birth of the baby.
Blood concentration HbA1c | 2.5 years
  The difference in blood concentration of HbA1c at the end of intervention (gestational week 37) between the intervention group and the control group, measured at baseline (gestational week 12-14), and at several occasions until 2 years after the birth of the baby.
Blood concentration CRP | 2.5 years
  The difference in blood concentration of CRP at the end of intervention (gestational week 37) between the intervention group and the control group, measured at baseline (gestational week 12-14), and at several occasions until 2 years after the birth of the baby.
Child body length | 2 years
  The difference in child body length (cm) between the intervention group and the control group, measured at baseline (birth), and at several occasions until 2 years after the birth of the baby.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual patient data due to limitations in ethical approval and data protection considerations of the project.